CLINICAL TRIAL: NCT03124108
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of Elafibranor at Doses of 80 mg and 120mg After 12 Weeks of Treatment in Patients With Primary Biliary Cholangitis and Inadequate Response to Ursodeoxycholic Acid
Brief Title: Study to Evaluate the Efficacy and Safety of Elafibranor in Patients With Primary Biliary Cholangitis (PBC) and Inadequate Response to Ursodeoxycholic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505B-216-1; 2016-003817-80 (EudraCT Number)
Record Dates: First submitted 2017-03-28; First posted 2017-04-21 (Actual); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Primary Biliary Cholangitis (PBC)
Keywords: Elafibranor; Primary Biliary Cholangitis; Alkaline phosphatase
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Study subjects will take two tablets per day orally before breakfast with a glass of water each morning
  Interventions: Drug: Placebo
- Elafibranor 80 mg (Active Comparator): Study subjects will take two tablets per day orally before breakfast with a glass of water each morning
  Interventions: Drug: Elafibranor 80 mg
- Elafibranor 120 mg (Active Comparator): Study subjects will take two tablets per day orally before breakfast with a glass of water each morning
  Interventions: Drug: Elafibranor 120 mg

INTERVENTIONS:
Drug: Elafibranor 80 mg — Two coated tablets daily for 12 weeks
  Other Names: GFT505
  Arms: Elafibranor 80 mg
Drug: Elafibranor 120 mg — Two coated tablets daily for 12 weeks
  Other Names: GFT505
  Arms: Elafibranor 120 mg
Drug: Placebo — Two coated tablets daily for 12 weeks
  Arms: Placebo

SUMMARY:
The primary objective of the study is to compare the effect of daily oral administration of elafibranor 80mg and 120 mg on change in serum alkaline phosphatase (ALP) to that of placebo in patients with PBC and inadequate response to Ursodeoxycholic acid (UDCA).

ELIGIBILITY:
Inclusion Criteria:

1. Must have provided written informed consent
2. Definite or probable PBC diagnosis as demonstrated by the presence of at least 2 of the following 3 diagnostic factors:

   * History of elevated ALP levels for at least 6 months prior to Day 0 (randomization visit)
   * Positive Anti-Mitochondrial Antibodies (AMA) titers (> 1/40 on immunofluorescence or M2 positive by enzyme-linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies
   * Liver biopsy consistent with PBC
3. ALP >= 1.67x upper limit of normal (ULN)
4. Taking UDCA for at least 12 months (stable dose for ≥ 6 months) prior to screening visit
5. Contraception: Females participating in this study must be of non-childbearing potential or must be using highly efficient contraception for the full duration of the study and for 1 month after the end of treatment.

Exclusion Criteria:

1. History or presence of other concomitant liver diseases
2. Screening creatine phosphokinase (CPK) > upper limits of normal (ULN)
3. Screening alanine transaminase (ALT) or aspartate aminotransferase (AST) > 5 ULN
4. Screening total bilirubin > 2 ULN
5. Screening serum creatinine > 1.5 mg/dl
6. Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as patients with markers of kidney damage or estimated glomerular filtration rate [eGFR] of less than 60 mL/min/1.73 m^2).
7. Patients with moderate or severe hepatic impairment (defined as Child-Pugh B/C)
8. Platelet count <150 X 10^3/microliter
9. Albumin <3.5 g/dL
10. Presence of clinical complications of PBC or clinically significant hepatic decompensation
11. If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating
12. Known history of human immunodeficiency virus (HIV) infection
13. Medical conditions that may cause non-hepatic increases in ALP (e.g., Paget's disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Head, Study Director — Genfit
Locations (24):
- United States (13):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Schiff Center for Liver Diseases, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Research Institute, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Northwell Health Institution, Manhasset, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- Hopital Saint-Antoine, Paris, France
- Germany (3):
  - Clinic for Gastroenterology and Hepatology, Cologne
  - University Hospital Frankfurt, Frankfurt
  - Johannes Gutenberg University, Mainz
- Spain (2):
  - Liver Unit, University of Barcelona, Barcelona
  - Hospital De La Sant Creu St. Pau, Barcelona
- United Kingdom (5):
  - University of Birmingham Centre for Liver Research, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - The Royal Liverpool University Hospital, Liverpool
  - King's College Hospital, London
  - The Newcastle Upon Tyne Hosptials NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Derived] Schattenberg JM, Pares A, Kowdley KV, Heneghan MA, Caldwell S, Pratt D, Bonder A, Hirschfield GM, Levy C, Vierling J, Jones D, Tailleux A, Staels B, Megnien S, Hanf R, Magrez D, Birman P, Luketic V. A randomized placebo-controlled trial of elafibranor in patients with primary biliary cholangitis and incomplete response to UDCA. J Hepatol. 2021 Jun;74(6):1344-1354. doi: 10.1016/j.jhep.2021.01.013. Epub 2021 Jan 21. PMID 33484775

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 68 participants were screened, out of which 45 participants were randomized, 15 participants in each of the 3 treatment groups.
Groups:
- Elafibranor 80mg: Participants received elafibranor 80 milligram (mg) tablets orally once daily for 12 weeks.
- Elafibranor 120mg: Participants received elafibranor 120 mg tablets orally once daily for 12 weeks.
- Placebo: Participants received matching placebo tablets orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Started | 15 | 15 | 15
Completed | 15 | 14 | 15
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 11 | 34
  >=65 years | 2 | 5 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (8.7) | 60.4 (6.9) | 60.5 (8.6) | 59.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 14 | 43
  Male | 1 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5 | 10
  Not Hispanic or Latino | 12 | 13 | 10 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 15 | 15 | 14 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Serum Alkaline Phosphatase (ALP) Levels at Week 12 (Endpoint)
Description: Relative change from baseline is in serum ALP levels at Week 12 (endpoint) were reported. Relative change from baseline is defined as percentage (%) change from baseline to endpoint.
Time Frame: Baseline, Week 12 (Endpoint)
Population: The modified Intent-to-Treat (mITT) analysis set included all randomized participants who received at least one study drug dose with available baseline value and at least one post baseline value for the primary endpoint.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percent change | -48.264 (14.7676) | -40.640 (17.3624) | 3.190 (14.8059)
Statistical Analysis 1: Comparison: Elafibranor 80mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference in percentage = -52.0, 95% CI 2-sided [-62.5 to -41.5], Standard Error of Mean 5.4
Statistical Analysis 2: Comparison: Elafibranor 120mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference in percentage = -43.9, 95% CI 2-sided [-55.7 to -32.1], Standard Error of Mean 6

2. Secondary Outcome: Percentage of Participants With Response Defined by Composite Risk Scores (ALP< 1.67 * Upper Limit of Normal [ULN] at Endpoint, Total Bilirubin [BIL] Within Normal Limits at Endpoint, and Greater Than [>] 15% ALP Reduction From Baseline to Endpoint)
Description: Percentage of participants with response defined by Composite Risk Scores (ALP Less than [<] 1.67 * ULN at endpoint, Total BIL within normal limits at endpoint, and > 15% ALP reduction from baseline to Endpoint) was reported.
Time Frame: Up to Week 12 (Endpoint)
Population: The mITT analysis set included all randomized participants who received at least one study drug dose with available baseline value and at least one post baseline value for the primary endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 66.7 | 78.6 | 6.7

3. Secondary Outcome: Percentage of Participants With Response Defined by Composite Risk Scores (ALP < 2 * Upper Limit of Normal at Endpoint, Total Bilirubin Within Normal Limits at Endpoint, and > 40% ALP Reduction From Baseline to Endpoint)
Description: Percentage of participants with response defined by composite risk scores (ALP < 2 * ULN at endpoint, Total BIL within normal limits at endpoint, and > 40% ALP reduction from baseline to endpoint) was reported.
Time Frame: Up to Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 73.3 | 42.9 | 0

4. Secondary Outcome: Percentage of Participants With Response Based on PARIS I Risk Score at Endpoint
Description: Percentage of participants with response based on Paris I risk score was defined as ALP less than or equal to (<=) 3 * ULN and aspartate aminotransferase (AST) <= 2 * ULN and bilirubin within normal limits.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 80.0 | 78.6 | 53.3

5. Secondary Outcome: Percentage of Participants With Response Based on PARIS II Risk Score at Endpoint
Description: Percentage of participants with response based on Paris II risk score was defined as ALP <= 1.5 * ULN and AST <= 1.5 * ULN and bilirubin within normal limits.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 53.3 | 50.0 | 0

6. Secondary Outcome: Percentage of Participants With Response Based on Toronto I Risk Score at Endpoint
Description: Percentage of participants with response based on Toronto I risk score was defined as ALP <= 1.67 *ULN.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 66.7 | 78.6 | 6.7

7. Secondary Outcome: Percentage of Participants With Response Based on Toronto II Risk Score at Endpoint
Description: Percentage of participants with response based on Toronto II risk scores was defined as ALP <= 1.75 * ULN.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 66.7 | 78.6 | 6.7

8. Secondary Outcome: Median Percentage Risk as Assessed by United Kingdom-Primary Biliary Cholangitis (UK-PBC) Risk Total Score at Endpoint
Description: UK-PBC risk score at endpoint estimated that the median percentage risk that a participant treated with ursodeoxycholic acid (UDCA) will develop liver failure requiring liver transplant in 5, 10 and 15 years. UK-PBC score was calculated at each of the 3 survivor functions 1-baseline survival function^exp(0.0287854*[alpEPxuln-1.722136304] - 0.0422873*[{(altastEPxuln/10)^-1} - 8.675729006] + 1.4199 * [ln{bilEPxuln /10}+2.709607778] -1.960303*[albxlln -1.17673001]-0.4161954*[ pltxlln -1.873564875]). Where: Baseline survivor function=0. 982 (at 5 years); 0. 941 (at 10 years); 0.893 (at 15 years). alpEPxuln = ALP at endpoint/upper level normal ALP; altastEPxuln=(ALT, AST) at endpoint/upper level normal of the value; bilEPxuln=bilirubin at endpoint/upper level normal bilirubin; albxlln=albumin at baseline/albumin lower level normal; pltxlln=platelet count at baseline/ platelet count lower level normal.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Median (Full Range); unit: Percentage risk
Groups:
- Elafibranor 120 mg: Participants received orally a dose of 120 mg elafibranor as tablets once daily for 12 weeks.
Arm/Group | Elafibranor 80mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage risk
  5 year risk at Week 12 | 0.80 [0.1 to 6.0] | 0.95 [0.2 to 5.8] | 1.30 [0.1 to 3.7]
  10 year risk at Week 12 | 2.60 [0.3 to 18.8] | 3.05 [0.8 to 18.1] | 4.40 [0.5 to 12.0]
  15 year risk at Week 12 | 4.70 [0.6 to 32.1] | 5.55 [1.5 to 31.0] | 8.00 [0.9 to 21.1]

9. Secondary Outcome: Percentage of Participants With Response Defined by 10, 20 and 40 Percent Reduction in Alkaline Phosphatase
Description: Percentage of participants with response (defined by at least 10%, 20%, and 40% decrease in ALP from baseline to Endpoint) reported.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- Elafibranor 80 mg: Participants received orally a dose of 80 milligram (mg) elafibranor as tablets once daily for 12 weeks.
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants
  10 Percent Reduction | 93.3 | 92.9 | 13.3
  20 Percent Reduction | 93.3 | 92.9 | 6.7
  40 Percent Reduction | 86.7 | 57.1 | 0

10. Secondary Outcome: Percentage of Participants With Response Defined by Normalized Alkaline Phosphatase Levels at Endpoint
Description: The response was defined by normalized ALP levels (ALP ULN 105 units per liter [U/L] for females, 129 U/L for males) at endpoint.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 13.3 | 21.4 | 0

11. Secondary Outcome: Percentage of Participants With Response Defined by Normalized Bilirubin (BIL) at Endpoint
Description: The response was defined by normalized BIL levels (BIL ULN <1.20 milligram per deciliter [mg/dL]) at endpoint.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 86.7 | 92.9 | 93.3

12. Secondary Outcome: Percentage of Participants With Response Defined by Normalized Albumin (ALB) Levels at Endpoint
Description: The response was defined by normalized ALB levels (3.5-5.2 gram per deciliter [g/dL] for ages 18-60 years; 3.2-4.6 g/dL for ages 61-91 years) at endpoint.
Time Frame: At Week 12 (Endpoint)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Percentage of participants | 100 | 100 | 100

13. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) Levels at Endpoint
Description: Change from baseline in ALT levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
U/L | -0.5 (57.38) | 7.3 (29.13) | -1.2 (8.57)

14. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) Levels at Endpoint
Description: Change from baseline in AST levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
U/L | 6.0 (55.29) | 11.1 (27.96) | -4.3 (7.97)

15. Secondary Outcome: Change From Baseline in Gamma-glutamyl Transferase (GGT) Levels at Endpoint
Description: Change from baseline in GGT levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
U/L | -91.5 (95.30) | -61.9 (70.82) | 0.6 (54.40)

16. Secondary Outcome: Change From Baseline in 5 Prime (') Nucleotidase Levels at Endpoint
Description: Change from baseline in 5' nucleotidase levels at endpoint was reported. 5' nucleotidase is an enzyme used as a biomarker of hepatobiliary cholestasis and is less sensitive but more specific than GGT and ALP.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
U/L | -7.81 (8.279) | -4.59 (13.067) | -0.47 (3.491)

17. Secondary Outcome: Change From Baseline in Total Bilirubin (BIL) Levels at Endpoint
Description: Change from baseline in total BIL levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
micromole per liter (mcmol/L) | -0.23 (3.425) | -0.51 (2.821) | -0.01 (3.548)

18. Secondary Outcome: Change From Baseline in Conjugated Bilirubin Levels at Endpoint
Description: Change from baseline in conjugated bilirubin levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
mcmol/L | 0.34 (2.229) | -0.06 (0.596) | 0.45 (1.526)

19. Secondary Outcome: Change From Baseline in Albumin Levels at Endpoint
Description: Change from baseline in albumin levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
gram per liter (g/L) | 2.2 (2.54) | 2.3 (2.73) | 0.0 (2.20)

20. Secondary Outcome: Change From Baseline in Cholesterol Levels at Endpoint
Description: Change from baseline in cholesterol levels at endpoints was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
millimole per liter (mmol/L) | -0.455 (0.7479) | -0.387 (0.6308) | 0.043 (0.3706)

21. Secondary Outcome: Change From Baseline in Low-density Lipoprotein (LDL) Cholesterol Levels at Endpoint
Description: Change from baseline in LDL-cholesterol at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
mmol/L | -0.366 (0.5919) | -0.334 (0.4848) | 0.061 (0.3272)

22. Secondary Outcome: Change From Baseline in High-density Lipoprotein (HDL) Cholesterol Levels at Endpoint
Description: Change from baseline in HDL-cholesterol levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
mmol/L | -0.017 (0.3898) | 0.059 (0.3391) | -0.007 (0.2988)

23. Secondary Outcome: Change From Baseline in Triglycerides Levels at Endpoint
Description: Change from baseline in triglycerides levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
mmol/L | -0.155 (0.3460) | -0.253 (0.2085) | -0.019 (0.3776)

24. Secondary Outcome: Change From Baseline in Total Free Bile Acid Levels at Endpoint
Description: Change from baseline in total free bile acid levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^-9 mole per liter (mol/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
10^-9 mole per liter (mol/L) | -248.88 (2496.672) | -673.71 (2962.097) | -135.20 (6777.727)

25. Secondary Outcome: Change From Baseline in Total Conjugated Bile Acid Levels at Endpoint
Description: Change from baseline in total conjugated bile acid levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^-9 mol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
10^-9 mol/L | 5008.99 (17844.304) | -3280.16 (10941.769) | 1873.22 (21795.349)

26. Secondary Outcome: Change From Baseline in Total Bile Acid Levels at Endpoint
Description: Change from baseline in total bile acid levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^-9 mol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
10^-9 mol/L | 4760.11 (18919.661) | -3953.86 (12008.620) | 1738.02 (26521.746)

27. Secondary Outcome: Change From Baseline in 7 Alpha-hydroxy-4-cholesten-3-one Levels at Endpoint
Description: Change from baseline in 7 alpha-hydroxy-4-cholesten-3-one levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^-9 mol/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
10^-9 mol/L | -16.29 (27.584) | -10.04 (28.606) | 5.22 (10.848)

28. Secondary Outcome: Change From Baseline in Fibroblast Growth Factor-19 Levels at Endpoint
Description: Change from baseline in fibroblast growth factor-19 levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
nanogram per liter (ng/L) | -21.67 (52.588) | -16.96 (38.933) | -47.08 (69.560)

29. Secondary Outcome: Change From Baseline in Immunoglobulin M (IgM) Levels at Endpoint
Description: Change from baseline in IgM levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
g/L | -0.339 (0.5846) | -0.472 (0.5507) | -0.076 (0.7227)

30. Secondary Outcome: Change From Baseline in Tumor Necrosis Factor Levels at Endpoint
Description: Change from baseline in tumor necrosis factor levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
ng/L | 0.066 (0.7829) | 0.154 (1.1374) | 0.053 (0.8329)

31. Secondary Outcome: Change From Baseline in Transforming Growth Factor Beta Levels at Endpoint
Description: Change from baseline in transforming growth factor beta levels at endpoint was reported,
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
ng/L | 734.7 (2103.75) | 297.2 (2762.61) | -1163.0 (4295.49)

32. Secondary Outcome: Change From Baseline in Interleukin 6 Levels at Endpoint
Description: Change from baseline in interleukin 6 levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
ng/L | -0.021 (0.8337) | -0.261 (0.5213) | -0.165 (0.5624)

33. Secondary Outcome: Change From Baseline in Plasminogen Activator Inhibitor-1 Antigen (AG) Levels at Endpoint
Description: Change from baseline in plasminogen activator inhibitor-1 AG levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
microgram per liter (mcg/L) | -0.483 (2.9839) | -1.739 (4.6587) | -1.456 (4.6448)

34. Secondary Outcome: Change From Baseline in Cytokeratin-18 Levels at Endpoint
Description: Change from baseline in cytokeratin-18 (M30 and M65) levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
picomole per liter (pmol/L)
  Cytokeratin-18 M30 | 26.12 (472.247) | 163.33 (499.500) | 17.93 (307.531)
  Cytokeratin-18 M65 | 114.31 (627.068) | 238.97 (611.520) | -53.16 (131.934)

35. Secondary Outcome: Change From Baseline in Autotaxin Levels at Endpoint
Description: Change from baseline in autotaxin levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
mcg/L | 4.6 (156.92) | 49.9 (77.25) | 35.1 (161.58)

36. Secondary Outcome: C-reactive Protein Level at Endpoint
Description: C-reactive protein level at endpoint was reported.
Time Frame: Week 12 (Endpoint)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: milligram per liter (mg/L)
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
milligram per liter (mg/L) | 2.74 [1.81 to 4.14] | 2.84 [1.68 to 4.78] | 4.01 [2.52 to 6.37]

37. Secondary Outcome: Change From Baseline in Haptoglobin Levels at Endpoint
Description: Change from baseline in haptoglobin levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
g/L | -0.265 (0.4271) | -0.254 (0.1088) | 0.025 (0.2244)

38. Secondary Outcome: Change From Baseline in Fibrinogen Levels at Endpoint
Description: Change from baseline in fibrinogen levels at endpoint was reported.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
g/L | -0.865 (0.9472) | -0.452 (0.5780) | -0.072 (1.0936)

39. Secondary Outcome: Change From Baseline in 5D-Itch Scale Total Score
Description: 5 dimensional (5D)-Itch Scale is a reliable, multidimensional measure of itching that has been validated in participants with chronic pruritus to detect changes over time. It consists of 5 domains: duration, degree, direction, disability, and distribution. The duration, degree and direction domains each include one item, while the disability domain has four items (sleep, leisure/social, housework/errands, work/school). All items of the first four domains were measured on a 5-point Likert scale. The distribution domain included 16 potential locations of itch, including 15 body part items (head/scalp, soles, face, palms, chest, abdomen, back, buttocks, thighs, lower legs, tops of feet/toes, tops of hands/fingers, upper arms, groin, forearms) and one point of contact with clothing or bandages. Scores of each of five domains are achieved separately and then summed together to obtain a total 5-D score. 5-D scores can potentially range between 5 (no pruritus) and 25 (most severe pruritus).
Time Frame: Baseline, Week 12 (Endpoint)
Population: The mITT analysis set included all randomized participants who received at least one study drug dose with available baseline value and at least one post baseline value for the primary endpoint. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 12 | 15
Units on a scale | -2.1 (5.15) | -0.1 (2.19) | 0.8 (4.93)

40. Secondary Outcome: Change From Baseline in Pruritus as Assessed by Visual Analogue Scale (VAS) Total Score
Description: The VAS is a reliable and validated method of pruritus assessment. The VAS is adequate in assessing the severity of the symptom; it does not take into account other aspects of pruritus, such as the relative impact of pruritus on quality of life. The VAS, for pruritus assessment, requires the participant to use abstract thought processes to convert their itch severity to a mark on a continuum. A participant draws a line anywhere on the scale ranging from 0 to 10 (where 0 represents 'no itching' and 10 represents 'worst possible itching') that best represents the severity of participant's itching and the scoring involves manual measuring of the mark with a ruler on range of 0 to 100 millimeter (mm). Higher scores indicate worse itching.
Time Frame: Baseline, Week 12 (Endpoint)
Population: The mITT analysis set included all randomized participants who received at least one study drug dose with available baseline value and at least one post baseline value for the primary endpoint. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 14 | 14 | 15
Units on a scale | -4.4 (22.80) | -4.7 (11.81) | 9.3 (35.93)

41. Secondary Outcome: Change From Baseline in Primary Biliary Cholangitis -40 (PBC-40) Quality of Life (QoL) Questionnaire Scores
Description: PBC-40 QoL Questionnaire is a patient-derived, disease-specific QoL measure developed and validated for use in PBC. It consists of 9 domains with total 40 questions as: 1) digestion and diet (questions 1-3, total score range: 3-15); 2) experiences (questions 4-7, total score range: 4-20); 3) itching (questions 8-10, total score range: 3-15); 4) fatigue (questions 11-18, total score range: 8-40); 5) effort and planning (questions 19-21, total score range: 3-15); 6) memory and concentration (questions 22-27, total score range: 6-30); 7) affects you as a person (questions 28-33, total score range: 6-30); 8) affects your social life (questions 34-37, total score range: 4-20); 9) overall impact on your life (questions 38-40, total score range: 3-15). PBC-40 QoL Questionnaire has 40 questions, each scored on scale of 1-5 (1 = least impact, 5 = greatest impact). For each domain, scoring involved summing individual question response scores. Higher scores indicate poorer quality of life.
Time Frame: Baseline, Week 12 (Endpoint)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Elafibranor 80 mg | Elafibranor 120 mg | Placebo
Number analyzed (Participants) | 15 | 14 | 15
Units on a scale
  Digestion and Diet | -0.3 (2.74) | -0.6 (2.24) | -0.6 (3.00)
  Experiences | 0.6 (2.64) | -1.3 (1.77) | -0.7 (3.69)
  Itching | -0.9 (6.19) | -4.1 (6.56) | 2.1 (5.78)
  Fatigue | -1.9 (4.10) | -1.4 (2.71) | -1.5 (5.04)
  Effort and Planning | -0.9 (2.03) | -0.8 (1.31) | -0.9 (1.98)
  Memory and concentration | 0.1 (3.26) | -1.5 (3.33) | -0.5 (3.25)
  Affecting you as a Person | -1.8 (3.78) | -2.5 (2.85) | -1.3 (3.22)
  Affects your Social Life | 1.3 (3.08) | 0.0 (1.47) | 1.4 (4.79)
  Impact on your Life | -0.1 (3.04) | 0.6 (0.63) | -1.0 (3.30)

42. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Treatment Emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical (investigational) product and which does not necessarily have to have a causal relationship with this treatment. A Serious adverse event (SAE) is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization/prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is another medically important condition. TEAEs is defined as (1) it is not present when active phase of study (time of first dose) begins and is not a chronic condition that is part of patient's medical history, or it is present at start of active phase or as part of patient's medical history, but severity/frequency increases during active phase.
Time Frame: Up to Week 12
Population: The Safety Set included all randomized participants who were administered at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
Number analyzed (Participants) | 15 | 15 | 15
Participants
  TEAEs | 12 | 13 | 12
  Serious TEAEs | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 16 Weeks
Arm/Group | Elafibranor 80mg | Elafibranor 120mg | Placebo
All-Cause Mortality (participants affected / at risk) | 13/15 | 13/15 | 12/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15 | 0/15
Other Adverse Events (participants affected / at risk) | 12/15 | 13/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elafibranor 80mg (N=15) | Elafibranor 120mg (N=15) | Placebo (N=15)
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elafibranor 80mg (N=15) | Elafibranor 120mg (N=15) | Placebo (N=15)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleral Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Cholesterol Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Urine Present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cystoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver Palpable (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine Albumin/Creatinine Ratio Increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Urobilinogen Urine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White Blood Cells Urine (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral Amyloid Angiopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nitrituria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 2 (3)
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stent Removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor retains exclusive ownership of all data, results, reports, findings, discoveries, and any other information collected during this study; these may not be published, given, or disclosed, either in part or in whole, by the Investigator or by any person under his/her authority to any third party without the prior express consent of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03124108/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT03124108/SAP_001.pdf